## Circulating tumour cells as biomarkers to predict prostate cancer metastasis for treatment stratification of localised cancer (C-ProMeta-1) CONSENT FORM

If you agree to the statement in the box, please indicate by writing your <u>initials</u>. If you do not agree please add 'X' in the box.

Please include initial or 'X'

| I confirm that I have read and understood the 'C-ProMeta-1 Patient Information Sheet' version 1 31/08/2021 and have had the content explained to me in sufficient detail. I have had an opportunity to ask questions and have had them answered satisfactorily. | | | |
|---|---|---|---|
| I consent to donate <u>additional blood samples</u> for rese follow up during my routine visits | | | |
| I understand that I may be contacted by the research team annually over a 10 year period as described in the patient information sheet version 1 31/08/2021 to gather information regarding my cancer recurrence and progression, my blood test results and further treatment. | | | |
| I consent to the Robert Lane Tissue Bank (RLTB) inc<br>specifically for current and future research purposes. | | | |
| I consent to my personal, identifiable and associated clinical information (from my medical records inclusive of imaging data), relevant to this condition, being stored indefinitely and securely and to be accessed by authorised staff in future to derive information about my health for research purposes. All staff undertaking current and future research will abide by the Data Protection Act 2018 UK with the reference to the General Data Protection Regulation (GDPR), or equivalent law in their respective jurisdiction. | | | |
| I agree that my blood derivatives and associated clinical information can be supplied in an anonymised form to non-profit organisations (i.e. NHS, Universities), commercial organisations or researchers involved in the commercial | | | |
| sector providing the purpose of the intended researc managing committee and the RLTB steering commit | | | |
| I agree that my blood derivatives and associated clinical information may be exported in an anonymised form outside of England, Wales, Northern Ireland providing the purpose of the intended research is to improve patient care, and has been approved by the study managing committee and the RLTB steering committee. | | | |
| I understand that I will not financially gain from donating my tissue or associated clinical information. These will not be sold. | | | |
| I agree that my samples, including my DNA and RNA, may be used in genetic research aimed at understanding the genetic influences on prostate cancer, but will not be released for research involving inherited disease and reproductive cloning. | | | |
| I understand that I am free to withdraw my consent at any time, without giving reason, and this will not affect my clinical care or legal rights. Upon withdrawing my consent, I have the option of requesting that my unprocessed blood and associated data, are disposed appropriately as per policy of sponsor and GDPR. | | | |
| Name of patient: | Date: | Signature: | MRN number: |
| | | | Date of Birth: |
| Name of person taking consent: | Date: | Signature: | Patient tracking no: |

For any further information or to withdraw consent, please contact: the study team by <a href="mailto:bci-cmetapro1@qmul.ac.uk">bci-cmetapro1@qmul.ac.uk</a> or Robert Lane <a href="mailto:Tissue Bank">Tissue Bank</a>, <a href="mailto:Centre for Biomarker and Biotherapeutics">Centre for Biomarker and Biotherapeutics</a>, <a href="mailto:Barts">Barts</a></a>
<a href="mailto:Cancer Institute">Cancer Institute</a>, <a href="mailto:Joseph Rotblat Building</a>, <a href="mailto:Charterhouse square">Charterhouse square</a>, <a href="mailto:London">London</a>, <a href="mailto:EC1M 6BQ">EC1M 6BQ</a> or <a href="mailto:020 7882 3739</a>

VERSION 1 31/08/2021 1